CLINICAL TRIAL: NCT05721300
Title: Study on Screening, Verification and Intervention of High-risk Patients With Liver Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Hospital (Xiamen), Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhongshanXiamenH-ZHB
Record Dates: First submitted 2022-12-22; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma; Chronic Hepatitis B
Keywords: Chronic hepatitis B (CHB); hepatocellular carcinoma (HCC); nucleos(t)ide analogues (NAs); interferon
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experience group (Experimental): patients receive NAs（"Entecavir"or"Tenofovir"or"Tenofovir alafenamide"） combine with interferon treatments for 48weeks, and then continue NAs treatment
  Interventions: Drug: NAs（"Entecavir"or"Tenofovir"or"Tenofovir alafenamide"） combined with interferon treatments
- control group (Active Comparator): patients receive NAs treatment（"Entecavir"or"Tenofovir"or"Tenofovir alafenamide"）
  Interventions: Drug: NAs （"Entecavir"or"Tenofovir"or"Tenofovir alafenamide"） treatments

INTERVENTIONS:
Drug: NAs（"Entecavir"or"Tenofovir"or"Tenofovir alafenamide"） combined with interferon treatments — NAs（"Entecavir"or"Tenofovir"or"Tenofovir alafenamide"） combine with interferon treatments for 48 weeks, and then continue with NAs treatment（"Entecavir"or"Tenofovir"or"Tenofovir alafenamide"）
  Other Names: IFN group
  Arms: experience group
Drug: NAs （"Entecavir"or"Tenofovir"or"Tenofovir alafenamide"） treatments — patients receive NAs（"Entecavir"or"Tenofovir"or"Tenofovir alafenamide"） treatment at least 48 weeks
  Arms: control group

SUMMARY:
The goal of this clinical trial is to test the outcomes of HBsAg(+) patients in the treatments of NAs vs NAs plus IFN . The main questions it aims to answer are:

1. Clinical effect analysis of nucleoside analogs (NAs) group a group and NAs plus interferon group after 48 weeks of treatment;
2. Repetitive effect and time effect of different drug treatment at different follow-up time points;
3. To evaluate the difference of therapeutic effect of NAs or NAs combined with interferon;
4. Follow up and compare the incidence of early liver cancer in each group. Participants will be asked to receive NAs or NAs combined with interferon treatments, and Regular blood sampling and color ultrasound examination.

Researchers will compare control group to see if occurrence of liver cancer.

ELIGIBILITY:
Inclusion Criteria (if one of them is met, it will be included):

1. HBsAg positive patients without liver cirrhosis:

1. Chronic hepatitis B virus（HBV） infected persons with positive serum HBV-DNA, if their alanine aminotransferase(ALT) continues to be abnormal and other causes of ALT increase are excluded;
2. In patients with positive serum HBV-DNA and normal ALT, liver histology showed obvious liver inflammation (≥ G2) or fibrosis (≥S2);
3. ALT continues to be normal (once every 3 months, lasting for 12 months), but there is a family history of cirrhosis/liver cancer and the age is>30 years old;
4. ALT is continuously normal (once every 3 months, lasting for 12 months), there is no family history of liver cirrhosis/liver cancer but the age is more than 30 years old, fibroscan or liver histology shows obvious liver inflammation or fibrosis;
5. Chronic HBV infected persons with negative serum HBV DNA who are receiving NA treatment or who have previously received NA treatment.

2. HBsAg positive with iver cirrhosis patients Patients with compensatory cirrhosis, regardless of ALT or HBeAg status. The diagnosis of hepatitis B cirrhosis is in accordance with the diagnostic criteria of Chronic Hepatitis B (2019). It shall conform to the following (1) and (2) (pathological diagnosis), or (1) and (3) (clinical diagnosis).

1. At present, HBsAg is positive, or HBsAg is negative, HBcAb is positive, and there is a clear history of chronic HBV infection (HBsAg positive in the past>6 months), excluding other causes.
2. Pathology of liver biopsy was consistent with liver cirrhosis.
3. two or more of the following 5 items are met, and non cirrhotic portal hypertension is excluded: ① Imaging examination shows signs of cirrhosis and (or) portal hypertension; ② Endoscopy showed esophageal and gastric varices; ③ The determination of liver hardness is consistent with liver cirrhosis; ④ Blood biochemical examination showed that the albumin level decreased (<35g/L) and/or prothrombin time（PT） prolonged (>3s longer than the control); ⑤ Blood routine examination showed that platelet count was<100 * 10 ^ 9/L.

Exclusion Criteria:(if one of them is met, it will be excluded)

1. Previous history of decompensated liver function or clinical symptoms of decompensated liver disease at baseline, such as hepatic encephalopathy, esophageal variceal bleeding, ascites, splenomegaly, etc.
2. In the first 6 months of screening, they received NA (such as lamivudine, adefovir dipivoxil tablets) or interferon treatment with high drug resistance rate;
3. Have received immunosuppressive agents or other immunomodulators (such as thymosin), systemic cytotoxic drugs, and effective antiviral therapy including Chinese herbal medicine (such as ganciclovir, lobcavir, and valaciclovir) within 6 months before screening.
4. The laboratory examination showed liver failure during screening.
5. There are evidences supporting the diagnosis of hepatocellular carcinoma, such as suspicious lesions found by ultrasound or imaging and/or serum alpha-fetoprotein (AFP)>50ug/L.
6. It is accompanied by hepatitis C virus（HCV）, hepatitis D virus （HDV） and HIV infection.
7. Presence of other liver diseases: combined with other pathogen infection, drug-induced liver injury, alcoholic hepatitis, nonalcoholic steatohepatitis, autoimmune liver disease, systemic diseases involving the liver, etc;
8. Subjects have other serious or active psychosomatic diseases, which may affect patients' treatment, evaluation or compliance with the study protocol. It includes any uncontrolled kidney, heart, lung, vascular, neurological, digestive, metabolic diseases (diabetes, thyroid and adrenal diseases), immune deficiency diseases or tumors with clinical significance.
9. There are contraindications to interferon treatment. Absolute contraindications include pregnancy, psychiatric history, uncontrolled epilepsy, decompensated cirrhosis, uncontrolled autoimmune disease, severe infection, retinal disease, heart failure, chronic obstructive pulmonary disease and other basic diseases. Relative contraindications include thyroid disease, past depression, uncontrolled diabetes, hypertension, and heart disease.
10. Have a history of allergy to nucleoside analogues.
11. The researchers believed that the compliance of the subjects was poor.
12. The researcher believes that the subject is not suitable to participate in this study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2215 (Estimated)
Dates: Start 2023-02-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of early liver cancer | 1-3 years
  To compare the incidence of early liver cancer in different treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: boheng zhang, Study Chair — Zhongshan Hospital (Xiamen), Fudan University
Locations (1):
- Boheng Zhang, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No